CLINICAL TRIAL: NCT04443322
Title: Safety and Efficacy Study of Durvalumab in Combination With Lenvatinib in Participants With Locally Advanced and Metastatic Hepatocellular Carcinoma-- DULECT2020-1 Trial
Brief Title: Durvalumab and Lenvatinib in Participants With Locally Advanced and Metastatic Hepatocellular Carcinoma ( Dulect2020-1 )
Acronym: Dulect2020-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RenJi-IIT-2020-0006
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-06

CONDITIONS: Liver Carcinoma; Liver Transplant; Complications
Keywords: liver cancer; liver transplant
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — durvalumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab and Lenvatinib (Experimental): Participants receive intravenous (IV) durvalumab at 1500mg on Day 1 of each 28-day cycle. Number of cycles: until unacceptable toxicity develops or >42 days before liver transplantation (If patients with locally advanced HCC would undergo liver transplant).
  Patients receive Lenvatinib 8-12mg(basing on weight), once a day, oral at least 38 days of each 6 weeks cycle until >7 days before liver transplantation(If patients with locally advanced HCC would undergo liver transplant).
  Interventions: Drug: Durvalumab Injection; Drug: Lenvatinib 4 MG

INTERVENTIONS:
Drug: Durvalumab Injection — Anti-PD-L1 Monoclonal Antibody
  Other Names: Durvalumab; Imfinzi
Drug: Lenvatinib 4 MG — Lenvatinib (Lenvima, Eisai China) is a novel angiogenesis inhibitor which targets vascular endothelial growth factor 1-3, fibroblast growth factor receptor 1-4, platelet-derived growth factor receptor β etc.
  Other Names: Lenvima

SUMMARY:
This study will evaluate the safety and efficacy of durvalumab in combination with lenvatinib in participants with locally advanced hepatocellular carcinoma before liver transplant and metastatic unresectable HCC.The primary hypothesis of this study are that patients with locally advanced HCC could benefit from durvalumab plus lenvatinib before liver transplant; patients with metastatic unresectable HCC could also benefit from durvalumab plus lenvatinib with respect to: 1)Progression Free Survival (PFS) ; or recurrence-free survival (RFS) if patients with locally advanced HCC underwent liver transplant; 2) Objective Response Rate (ORR); and 3) Overall survival (OS). The investigators design a clinical study to explore whether the combination above as a treatment in patients with advanced and recurrent endometrial carcinoma could prolong PFS and to analyze potential immune biomarker of therapeutic response.

DETAILED DESCRIPTION:
The combination of Lenvatinib and Programmed death-ligand 1 (PD-L1) blocking has great potential in the treatment of locally advanced hepatocellular carcinoma before liver transplant and metastatic unresectable HCC. This trial is designed as a prospective, open label study for 20 patients with locally advanced hepatocellular carcinoma before liver transplant and metastatic unresectable HCC. The aim is to investigate the efficacy of the combination therapy of Lenvatinib 80-120mg daily orally and durvalumab 1500mg by IV infusion every 4 weeks in terms of progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically or by radiological criteria proven hepatocellular carcinoma; known mixed histology (e.g. hepatocellular carcinoma plus cholangiocarcinoma) or fibrolamellar variant is not allowed
* Locally advanced and metastatic HCC
* Has an eligibility scan (CT of the chest, triphasic CT scan or MRI of the abdomen, and CT or MRI of the pelvis) <1 week before the treatment of durvalumab in combination with lenvatinib.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to Cycle 1, Day 1.
* Has a Child-Pugh A liver score (5 to 6 points) within 7 days prior to Cycle1, Day 1.
* Has controlled hepatitis B (Hep B)
* The estimate time length between enrollment and liver transplantation should be at least 2 months
* No prior systemic therapy, local therapy (TACE etc.)>6w
* If female, is not pregnant or breastfeeding, and at least one of the following conditions applies: 1) Is not a woman of childbearing potential (WOCBP); or 2) Is a WOCBP and using a contraceptive method that is highly effective or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (a WOCBP must have a negative pregnancy test within 72 hours before the first dose of study treatment).
* Has adequate organ function.
* Granulocytes >= 1,500/uL
* Hemoglobin >= 8.5 g/dL; patients with recent or ongoing gastrointestinal bleed may not be transfused to reach the entry hemoglobin of 8.5 g/dL; physicians should ensure patients requiring transfusion prior to registration do not have an occult or clinically apparent gastrointestinal bleed
* Platelets >= 75,000/uL
* Creatinine =< 1.5 x upper limit of normal (ULN) (or creatinine clearance calculated >= 60 cc/minute)
* Bilirubin =< 3 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =<5 x ULN
* Prothrombin time (PT)-international normalized ratio (INR) =< 1.7 (not required for patients on anticoagulation agents; patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists)
* Patients with a history of hypertension should be well controlled (< 140/90 mmHg) on a regimen of anti-hypertensive therapy
* Significant history of cardiac disease is not allowed:
* Congestive heart failure > class II New York Heart Association (NYHA) Myocardial infarction within 6 months prior to registration Serious myocardial dysfunction, defined as scintigraphically (multigated acquisition scan [MUGA], myocardial scintigram) determined absolute left ventricular ejection fraction (LVEF) below 45% or an LVEF on echocardiogram(ECHO) below the normal limit at the individual institution

Exclusion Criteria:

* Has had esophageal or gastric variceal bleeding within the last 6 months.
* Has clinically apparent ascites on physical examination.
* Has had clinically diagnosed hepatic encephalopathy in the last 6 months.
* Has received local therapy to liver ablation other than with radiofrequency or microwave ablation.
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy.
* Has dual active Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) infection at study entry.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has known active tuberculosis (TB; Bacillus tuberculosis).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received prior systemic anti-cancer therapy for HCC including investigational agents.
* Is receiving any of the following prohibited concomitant therapies:1) Antineoplastic systemic chemotherapy or biological therapy; 2) Immunotherapy not specified in this protocol; 3) Investigational agents other than pembrolizumab; 4) Radiation therapy; 5) Oncological surgical therapy; or systemic glucocorticoids for any purpose other than to modulate symptoms from an AE that is suspected to have an immunologic etiology.
* Has received a live vaccine within 30 days prior to the first dose of study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to Cycle 1, Day 1.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Cycle 1, Day 1.
* Has severe hypersensitivity (≥Grade 3) to Durvalumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 3 years
  Defined as time from randomisation to first progression by investigator assessment using modified RECIST 1.1 or death (by any cause in the absence of progression)
Recurrence-Free Survival (RFS) | Up to 4 years
  If patients with locally advanced HCC would undergo liver transplant after neoadjuvant treatment of Durvalumab and Lenvatinib.RFS is defined as the time from randomization to first documentation of disease recurrence (local, regional, or distant) as assessed by BICR or by pathology consistent with HCC if required per the site's standard of care, or death due to any cause (both cancer and non-cancer causes of death)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 1 year
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.
Overall Survival (OS) | Up to 5 years
  Defined as the time from randomisation to death due to any cause
Percentage of Participants who Experience an Adverse Event (AE) | Up to 2 years
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-jun Zhang, MD, Study Director — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU; Qiang Xia, MD, Study Chair — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU; Hao Feng, MD., Ph.D., Principal Investigator — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China